CLINICAL TRIAL: NCT06005753
Title: Improving the Surgical Treatment of Injuries and Consequences of Injuries of the Acetabulum
Brief Title: Surgical Treatment of Injuries and Consequences of the Acetabulum
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Scientific Center of Traumatology and Orthopedics named after academician N.D. Batpenov (Other Government)
Responsible Party: Principal Investigator, Olzhas Bekarissov, Chief of NSCTO, National Scientific Center of Traumatology and Orthopedics named after academician N.D. Batpenov
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BR11065157(04)
Record Dates: First submitted 2023-08-15; First posted 2023-08-22 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Acetabular Fracture
Keywords: acetabulum; osteosynthesis; Stoppa approach; fracture
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group A (Experimental): Surgical intervention group
  Interventions: Procedure: Ostheosynthesis of acetabular fractures

INTERVENTIONS:
Procedure: Ostheosynthesis of acetabular fractures — The using of plate for fixation of acetabular fractures in surgical treatment

SUMMARY:
The aim of the program is to develop technologies for the diagnosis and treatment of injuries and consequences of the pelvis.

Purpose: to improve the technique of surgical treatment of acetabular fractures.

DETAILED DESCRIPTION:
Tasks: Implementation of low-traumatic access to the acetabulum; introduction of a new implant for osteosynthesis of complex acetabular fractures into clinical practice; мathematical modeling of fixation of the acetabulum with a new implant; рublication of the results of the work carried out The relevance of the use of new implants in orthopedics is due to the problem of adaptation of implants in the body, especially with poor quality of bone tissue. Currently, work is underway to improve the materials and shapes of implants, new alloys are being studied, polymer implants are being introduced, but the problem of their integration into bones remains. A promising direction in orthopedics is the creation of implants as close as possible in their morphological shape and elasto-strength properties to human bone. But the creation of an absolute copy of the bone structure from a metal alloy leads to a weakening of its strength and loss of fixation stability, and subsequent lysis of the adjacent bone tissue.

All this indicates the need for further search for new, perhaps more promising and effective ways to solve this problem.

ELIGIBILITY:
Inclusion Criteria:

* patients over 18 years of age
* patients with acetabular fractures undergoing surgery
* acetabular fractures according to the classification of Judet and Letournel

Exclusion Criteria:

* patients under 18 years of age
* posterior wall fracture according to the classification of Judet and Letournel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-11-25 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
consolidation of fracture | 1 year follow-up
  Evaluation of results using the radiological Matta criterion, the Harris Hip Score

CONTACTS AND LOCATIONS:
Locations (1):
- Center of National Scientific center Of Traumatology and Orthopedics named after academician N.D. Batpenov, Astana, Kazakhstan

IPD SHARING:
Plan to Share IPD: No